CLINICAL TRIAL: NCT05936671
Title: Quality of Recovery After Electroencephalogram and Nociception Level-guided Versus Standard Anesthesia Care in Female Patients Undergoing Laparoscopic Gynecological Surgery: A Randomized Controlled Trial
Brief Title: EEG and ANI Guided Anesthesia and Quality of Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3-2023-0116
Record Dates: First submitted 2023-06-13; First posted 2023-07-10 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Laparoscopic Gynecological Surgery
MeSH Terms: interventions — Sevoflurane; Remifentanil; Electroencephalography

STUDY DESIGN:
Intervention Model Description: Prospective, single-blinded, parallel-group, randomized clinical study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, medical staff who measure outcome variables, surgeons and nurses in the recovery room and wards are blinded so that medical staff and patients do not know the patient's assigned group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEG-and-ANI-guided group (Experimental): During anesthetic maintenance, sevoflurane concentration will be titrated according to EEG monitoring. Sevoflurane concentration will be titrated to maintain intraoperative Patient state index (PSi) ≥ 35 and to avoid burst suppression. Intraoperative target-controlled infusion of remifentanil will be titrated to maintain intraoperative ANI between 50 and 70.
  Interventions: Procedure: EEG-and-ANI-guided anesthesia; Drug: Sevoflurane and remifentanil; Device: EEG and ANI
- Usual care group (Active Comparator): During anesthetic maintenance, the attending anesthesiologists will provide a routine standard care for anesthetic and analgesic titration. In brief, hemodynamic variables and clinical situations will be used to titrate the sevoflurane concentration and remifentanil infusion rates.
  Interventions: Procedure: standard anesthesia; Drug: Sevoflurane and remifentanil

INTERVENTIONS:
Procedure: EEG-and-ANI-guided anesthesia — During anesthetic maintenance, sevoflurane concentration will be titrated according to EEG monitoring. Sevoflurane concentration will be titrated to maintain intraoperative Patient state index (PSi) ≥ 35 and to avoid burst suppression. Intraoperative target-controlled infusion of remifentanil will be titrated to maintain intraoperative ANI between 50 and 70.
  Arms: EEG-and-ANI-guided group
Procedure: standard anesthesia — During anesthetic maintenance, the attending anesthesiologists will provide a routine standard care for anesthetic and analgesic titration. In brief, hemodynamic variables and clinical situations will be used to titrate the sevoflurane concentration and remifentanil infusion rates.
  Arms: Usual care group
Drug: Sevoflurane and remifentanil — For anesthetic maintenance, balanced anesthesia with sevoflurane inhalation and target controlled infusion of remifentanil will be performed.
Device: EEG and ANI — EEG monitoring using SEDline (Masimo, Irvine, California, USA) and Analgesia Nociception Index (ANI; MetroDoloris Medical Systems, Lille, France) monitoring will be performed.
  Arms: EEG-and-ANI-guided group

SUMMARY:
This study aims to assess whether electroencephalogram (EEG) and nociception level-guided anesthesia can improve quality of recovery after laparoscopic gynecological surgery compared with standard care. Patients will be randomly assigned to either EEG and Analgesia Nociception Index (ANI)-guided anesthesia group (EEG-and-ANI-Guided group) or usual care group (control group). Primary outcome is 15-item Quality of Recovery (QoR-15) score at postoperative day (POD) 1. Secondary outcomes included remifentanil consumption during anesthesia, occurrence of awareness with recall, incidence of undesirable intraoperative movement, emergence time, postoperative pain scores, quality of recovery score at POD 2, and length of hospital stay.

DETAILED DESCRIPTION:
Adult women scheduled to undergo laparoscopic gynecologic surgery will be screened for eligibility. Patients will be randomly allocate to either the EEG-and-ANI-guided group or usual care group.

In the guided group, sevoflurane concentration will be titrated according to EEG monitoring. Intraoperative infusion of remifentanil will be titrated by ANI monitoring.

In the usual care group, EEG and ANI sensor will be attached to patients, but EEG and ANI monitor will be blinded to the attending anesthesiologists. The anesthesiologists will provide a standard care of our institution for anesthetic and analgesic titration. In brief, hemodynamic variables and clinical situations will be used to titrate the anesthetic depth and analgesic dose.

Blinded investigator will assess quality of recovery questionnaire-15 at postoperative day 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

Adult female patients who are scheduled to undergo laparoscopic gynecological surgery.

1. Total laparoscopic hysterectomy with/without salpingo-oophorectomy
2. Laparoscopic myomectomy
3. Laparoscope-guided salpingo-oophorectomy
4. Laparoscope-guided ovarian cystectomy
5. Laparoscope-guided enucleation of ovarian cyst

Exclusion Criteria:

1. Patients with nonregular sinus cardiac rhythm
2. Patients with implanted pacemakers
3. Patients on antimuscarinic agents, α2-adrenergic agonists, β1-adrenergic antagonists, antiarrhythmic agents
4. pregnant or breastfeeding women
5. Patients who are unable to communicate

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patient
Enrollment: 126 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-06-19 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
15-item Quality of Recovery (QoR-15) at postoperative day (POD) #1 | 24 hours after the end of surgery
  The Korean version of 15-item Quality of Recovery (QoR-15) score. Each item uses an 11-point numeric rating scale. The sum of the scores of the 15 items ranges from 0 to 150, with a high score indicating good quality of recovery.

SECONDARY OUTCOMES:
Remifentanil consumption during anesthesia | During surgery, from the anesthetic induction to emergence of anesthesia
  Total remifentanil consumption during anesthesia
Occurrence of awareness with recall | During the operation.
  Occurrence of awareness with recall during surgery, which will be asked at postoperative day #1.
Incidence of undesirable intraoperative movement | During the operation.
  Incidence of undesirable intraoperative movement during surgery
Intraoperative end-tidal sevoflurane minimum alveolar concentration (MAC) | During the operation
  Intraoperative end-tidal sevoflurane minimum alveolar concentration (MAC)
Intraoperative time ANI <50 [%] | During the operation.
  Intraoperative time of ANI value <50 / total duration of surgery (%)
Intraoperative mean PSi | During the operation.
  Intraoperative mean Patient state index (a processed EEG parameter related to a patient's current level of sedation/anesthesia along a scale of 0 to 100, where 100 represents being fully awake)
Intraoperative mean ANI | During the operation.
  Intraoperative mean Analgesia Nociception Index (expressed on a non-unit scale of 0-100; 100 indicates maximal relative parasympathetic tone)
Intraoperative EEG burst suppression | During the operation
  Intraoperative occurrence of burst suppression on electroencephalogram
burst suppression ratio | During the operation
  Intraoperative burst suppression ratio on electroencephalogram
burst suppression duration | During the operation
  duration of burst suppression on electroencephalogram
Emergence time | From time of administration of reversal agents of neuromuscular block until time of extubation, assessed up to 2 hours
  time between reversal of neuromuscular block and extubation
Intraoperative hypotension | During the operation
  Incidence of hypotension during surgery
Intraoperative phenylephrine consumption | During the operation.
  total dose of phenylephrine consumption during surgery
Pain numeric rating scale (NRS) | scores during post-anesthesia care unit (PACU) stay, at postoperative 24, 48 hours
  NRS (0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable ") pain scores during post-anesthesia care unit (PACU) stay, at postoperative 24, 48 hours
The incidence of post-operative nausea and vomiting | during the post-anesthesia care unit (PACU) stay, at postoperative day 1, 2
  The incidence of post-operative nausea and vomiting
Patient satisfaction with anesthetic management | At post-operative 24 hours
  Patient satisfaction with overall anesthetic management in 11-point scale (0-10), The higher the score, the higher the patient's satisfaction.
Quality of Recovery Questionnaire (15-item Quality of Recovery) at postoperative day #2 | At post-operative 48 hours
  Each item uses an 11-point numeric rating scale. The sum of the scores of the 15 items ranges from 0 to 150, with a high score indicating good quality of recovery.
shivering, airway obstruction, respiratory depression, sedation in PACU | from time of the post-anesthesia care unit (PACU) admission to time of discharge from PACU, assessed up to 2 hours
  Incidence of shivering, airway obstruction, respiratory depression, sedation
Hospital length of stay | From date of hospital admission until the date of hospital discharge, assessed up to 100 weeks
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Dong Woo Han, MD,PhD, Principal Investigator — Gangnam Severance Hospital
Locations (2):
- South Korea (2):
  - GangnamSeverance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul

REFERENCES:
- [Background] Punjasawadwong Y, Phongchiewboon A, Bunchungmongkol N. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD003843. doi: 10.1002/14651858.CD003843.pub3. PMID 24937564
- [Background] Upton HD, Ludbrook GL, Wing A, Sleigh JW. Intraoperative "Analgesia Nociception Index"-Guided Fentanyl Administration During Sevoflurane Anesthesia in Lumbar Discectomy and Laminectomy: A Randomized Clinical Trial. Anesth Analg. 2017 Jul;125(1):81-90. doi: 10.1213/ANE.0000000000001984. PMID 28598927
- [Background] Espitalier F, Idrissi M, Fortier A, Belanger ME, Carrara L, Dakhlallah S, Rivard C, Brulotte V, Zaphiratos V, Loubert C, Godin N, Fortier LP, Verdonck O, Richebe P. "Impact of Nociception Level (NOL) index intraoperative guidance of fentanyl administration on opioid consumption, postoperative pain scores and recovery in patients undergoing gynecological laparoscopic surgery. A randomized controlled trial". J Clin Anesth. 2021 Dec;75:110497. doi: 10.1016/j.jclinane.2021.110497. Epub 2021 Sep 28. PMID 34597955